CLINICAL TRIAL: NCT04323384
Title: The Effect of Biotene® Oralbalance Moisturizing Gel on the Symptoms of Xerostomia and the Efficiency and Ease of Mastication and Swallowing
Brief Title: The Effect of Biotene® on the Symptoms of Xerostomia and Mastication and Swallowing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Rebecca, Assistant Professor, Co-Primary Investigator, Nova Scotia Health Authority
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 23677
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Xerostomia; Hyposalivation
Keywords: swallowing; saliva; oral health; mastication; quality of life; artificial saliva
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Intervention Model Description: This project will use a crossover, repeated measures design to test the previously stated hypotheses. The benefits of using this design include improved control of between-subject variability and improved statistical power.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Biotene® followed by Sham (Experimental): Recruited volunteers will each participate in two experimental sessions. Participants will be randomized into either Protocol A or Protocol B. In their first session, participants in Protocol A will undergo baseline mastication, swallowing, salivary, and oral health-related quality of life testing, then they will receive the experimental condition. For the experimental condition, participants will be instructed to apply Biotene® Oralbalance Moisturizing Gel according to package directions. Testing will then be repeated. In the second session, after baseline testing, participants will receive the sham condition (instead of the experimental condition). For the sham condition, participants will be instructed to rinse their mouth with room temperature distilled water. Testing will then be repeated.
  Interventions: Device: Biotene® Oralbalance Moisturizing Gel
- Sham followed by Biotene® (Experimental): Recruited volunteers will each participate in two experimental sessions. Participants will be randomized into two protocols: 1) Protocol A and 2) Protocol B. In their first session, participants in Protocol B will undergo baseline mastication, swallowing, salivary, and oral health-related quality of life testing, then they will receive the sham condition. Testing will then be repeated. In the second session, after baseline testing, participants will receive the experimental condition (instead of the sham condition). Testing will then be repeated.
  Interventions: Device: Biotene® Oralbalance Moisturizing Gel

INTERVENTIONS:
Device: Biotene® Oralbalance Moisturizing Gel — Biotene® Oralbalance Moisturizing Gel will be applied to the oral cavity according to the package directions.

SUMMARY:
This study will compare the effects of Biotene® Oral Balance Moisturizing Gel (Biotene), an over-the-counter artificial saliva, that the effects of a sham condition on oral health-related quality of life, mastication, and swallowing in four groups of participants: 1) Participants not experiencing xerostomia or hyposalivation, 2) Participants experiencing xerostomia and hyposalivation, 3) Participants experiencing xerostomia but not hyposalivation, 4) Participants experiencing hyposalivation but not xerostomia.

DETAILED DESCRIPTION:
Saliva is important for maintaining oral and general health. This complex bioactive substance serves many functions including i) protecting the oral mucosa, ii) reducing demineralization and facilitating remineralization of teeth, and iii) sustaining a balanced oral biome and facilitating antimicrobial actions and clearance of pathogens. Moreover, saliva also plays a critical role in alimentary functions such as mastication and swallowing.

The role of saliva in the process of mastication and swallowing is complex and is not currently well understood. The purpose of mastication is to process food in the oral cavity into a bolus that can be transported through the oropharynx, swallowed safely, and then easily digested. During mastication, ingested food particles are mechanically reduced in size through the process of lingual particle selection and fragmentation between the occlusal surfaces of the teeth. The secretion of saliva is critical for effective mastication, bolus formation and bolus transport. There is also evidence to suggest that the volume of saliva secreted into the oral cavity during alimentation may impact swallowing biomechanics.

Oral tissue dryness is a complex issue. Hyposalivation and xerostomia span numerous clinical pathologies and are known side effects of many therapeutic agents. Hyposalivation occurs when there are objective signs of a reduction of the amount of saliva produced by the salivary glands and can be measured using sialometry. Xerostomia refers to the subjective symptoms of dry mouth and can only be assessed through a person's perception of the presence of symptoms. A person may experience xerostomia with or without hyposalivation or experience hyposalivation with or without xerostomia. Hyposalivation is a commonly complaint in older adults. Additionally, patients with hyposalivation and xerostomia frequently report symptoms of dysphagia, or difficulty swallowing.

To alleviate symptoms associated with hyposalivation, such as the perception of dry mouth, or xerostomia, many people use over-the-counter artificial saliva products such as Biotene® Oral Balance Moisturizing Gel (Biotene). There is, however, a paucity of evidence examining the effect of these products on oral health-related quality of life, mastication, and swallowing. The goal of this study therefore, is to compare the effects of Biotene® Oral Balance Moisturizing Gel (Biotene) with the effects of a sham condition on oral health-related quality of life, masticatory efficiency, and perceived swallowing effort in four groups of participants: 1) Participants not experiencing xerostomia or hyposalivation, 2) Participants experiencing xerostomia and hyposalivation, 3) Participants experiencing xerostomia but not hyposalivation, 4) Participants experiencing hyposalivation but not xerostomia.

It is hypothesized that, following the application of Biotene® Oralbalance Moisturizing Gel, all groups of participants will experience improved oral health-related quality of life, improved masticatory efficiency a reduction in perceived swallowing effort. The reduction will be significant when compared with that of the sham condition. Participants with xerostomia and/or hyposalivation will demonstrate greater improvement in oral health-related quality of life, improvement in masticatory efficiency, and reduction in perceived swallowing effort compared with those who do not experience xerostomia and/or hyposalivation.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable adults
* Age 19 years of age or older
* Able to sit upright independently and transfer to a chair
* Able to eat foods requiring mastication
* Decision-making capacity to provide informed consent

Exclusion Criteria:

* Acute illness or uncontrolled medical condition
* Allergies to any pharmaceuticals
* Allergies to medical tape/adhesive
* Allergies to Nabisco Saltines® or any of the ingredients
* Participant-reported issues with excess saliva and/or drooling
* Open ulcerations in the oral cavity.

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived Swallowing Effort after application of Biotene®/Sham | baseline, after application of Biotene®/sham
  Participants will be instructed to swallow and use a visual analog scale to rate the perceived swallowing effort by bisecting a 100mm line anchored with "no effort" and "extreme effort" (higher scores indicate a worse outcome). After the experimental or sham condition has been applied, participants will re-rate their perceived swallowing effort.

SECONDARY OUTCOMES:
Change in Spontaneous Swallowing Frequency after application of Biotene®/Sham | baseline, after application of the Biotene®/sham
  Spontaneous swallowing frequency will be derived from four physiologic signals. These include, simultaneous respiratory movements (swallowing apnea), surface movements associated with hyolaryngeal excursion recorded via a pressure pad transducer, and acoustic signals associated with hyolaryngeal excursion obtained using a contact microphone adhered to the skin just below the lateral cricoid cartilage, and event marking using an independent rater.
Change in the Test of Masticating and Swallowing Solids (TOMASS) after application of Biotene®/Sham | baseline, after application of the Biotene®/sham
  The TOMASS will be used to evaluate masticatory efficiency. Participants will be instructed to eat a single portion of a cracker "as quickly as is comfortably possible and when you have finished, say your name out loud". Two independent raters will observe a lateral view of the face and count masticatory cycles by observing jaw movements. Timing of the entire task will be recorded using a stopwatch. Longer mastication times/more masticatory cycles required to eat the cracker are a worse outcomes.
Change in the Effectiveness of Mastication and Swallowing after application of Biotene®/Sham | baseline, after application of the Biotene®/sham
  Effectiveness of mastication and swallowing will be measured based on cleansability of debris in the oral cavity. Pictures of the oral cavity will be taken before and after chewing the cracker and a score will be assigned based on the amount of residual cracker in the oral cavity. The criteria used to assign a rating (0-2) will be based on the Oral Health Assessment Tool (OHAT). Higher values indicate worse outcomes.
Change in Oral Health-Related Quality of Life after application of the Biotene®/sham | baseline, after application of the Biotene®/sham condition, half hour increments until responses revert to baseline
  A combination of the Oral Health Quality of Life Inventory (OH-QoL) survey and the Eight-item Visual Analogue Scale (VAS) xerostomia questionnaire will be used to measure oral health-related quality of life. Questions from the OH-QoL specific to moisture will be administered and participants will rate their responses on a likert scale (1=somewhat important; 2=very important), and to understand the effect Biotene® Oralbalance Moisturizing Gel on oral health quality of life, "How happy are you with how moist your mouth feels?" will be asked before and after the application of Biotene® Oralbalance Moisturizing Gel or the sham. The eight-item VAS xerostomia questionnaire will also be administered asked before and after the application of Biotene® Oralbalance Moisturizing Gel or the sham (higher scores indicate worse outcomes).

CONTACTS AND LOCATIONS:
Overall Officials: Leigha Rock, PhD, Principal Investigator — Nova Scotia Health Authority/Dalhousie University

IPD SHARING:
Plan to Share IPD: No